CLINICAL TRIAL: NCT06227039
Title: Using Augmented Reality With Vibroacoustic Stimulation to Improve the Patient Experience During In-Office Otorhinolaryngology Procedures
Brief Title: Patient Augmented Reality and Vibratory Array Otorhinolaryngology Procedures
Acronym: PARVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, James Daniero, MD, Associate Professor, Division Director, Laryngology and Voice Care, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSR210111
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pain, Acute; Vocal Fold Polyp; Vocal Cord Paralysis; Laryngeal Neoplasms
MeSH Terms: conditions — Acute Pain; Vocal Cord Paralysis; Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No treatment (No Intervention): This arm will be the current standard of care
- Vibroacoustic (Experimental): This arm will use the vibroacoustic device to provide a mechanical stimulus to the patient as treatment to reduce pain and anxiety. Augmented reality glasses will be worn but will be turned off.
  Interventions: Other: Vibroacoustic stimulation on; Other: Augmented reality off
- Augmented Reality (Experimental): This arm will use the augmented reality game to provide a visual stimulus to the patient as treatment to reduce pain and anxiety. Vibroacoustic device will be worn but will be turned off.
  Interventions: Other: Augmented Reality on; Other: Vibroacoustic stimulation off
- Combination vibroacoustic and augmented reality (Experimental): This arm will use both the augmented reality game and vibroacoustic device to provide a visual stimulus to the patient as treatment to reduce pain and anxiety.
  Interventions: Other: Vibroacoustic stimulation on; Other: Augmented Reality on

INTERVENTIONS:
Other: Vibroacoustic stimulation on — Mechanical stimulus is provided to the patient through a vibroacoustic device via vibration around the neck.
  Arms: Combination vibroacoustic and augmented reality; Vibroacoustic
Other: Augmented Reality on — Visual stimulus is provided through augmented reality glasses in the form of a game.
  Arms: Augmented Reality; Combination vibroacoustic and augmented reality
Other: Vibroacoustic stimulation off — Vibroacoustic device is worn but turned off.
  Arms: Augmented Reality
Other: Augmented reality off — Augmented reality glasses are worn but turned off.
  Arms: Vibroacoustic

SUMMARY:
In-office procedures (IOPs) are a cost-effective, and safe alternative to many operating room procedure, with benefits such as reduced anesthesia risk. One of the major causes of failed in-office procedures or requirement of conversion to the operating room is poor patient tolerance. Vibration and augmented reality (AR) can be used as non-pharmacologic treatment options to treat patient anxiety and pain by using the physiology proposed by the gate-way theory of pain as well as distraction. This study seeks to compare anxiety and pain perception with patient reported survey data, as well as physiologic indicators of stress such as heart rate variability (HRV) within patients undergoing IOPs in a laryngology office with and without vibration and AR treatment.

DETAILED DESCRIPTION:
In-office procedures (IOPs) represent a cost-effective and safe alternative to operating room procedures for a myriad of disease processes across medical and surgical specialties. IOPs are performed under local anesthetic without general anesthesia or sedation, resulting in faster and often safer procedures by eliminating risks associated with general anesthesia. IOPs are primarily limited by patient tolerance, as there is a lack of currently available non-pharmacologic treatment options for patient anxiety, stress, discomfort, and pain during these procedures.

The Gate Control Theory of Pain postulates that only a limited amount of simultaneous sensory stimuli can be processed by the central nervous system and therefore non-painful stimuli, such as vibration or virtual distraction (i.e. virtual or augmented reality), can eliminate or lessen the perception of concurrent painful stimuli. The use of these non-painful stimuli has been shown to have clinical utility in the setting of procedures such as percutaneous injections and wound dressing changes.

However, the coupling of multiple sensory distraction techniques has not been described for IOPs. Furthermore, no investigation of sensory distraction techniques to reduce patient discomfort within the field of otolaryngology has been conducted. The focus of the proposed project is to improve patient experience during IOPs by coupling a novel vibroacoustic stimulation device with original AR software applications.

In-office otolaryngology procedures specifically involve using a rigid endoscope or a flexible nasolarynogoscopy to visualize the inside of a patient nose, sinus, posterior oropharynx, and vocal cords. Using these imaging modalities, awake, in-office procedures can be performed. However, these procedures are often very uncomfortable and anxiety producing.

The goal of the study is to determine whether or not wearing an augmented reality headset with a novel game and vibroacoustic simulation device can help reduce anxiety and improve the patient experience of in-office otolaryngology procedures. The device consists of an augmented reality headset worn by the patient, a vibration device that is applied to the patient's neck to help reduce the sensation of the procedure, and a clicker that allows the patient to interact with the augmented reality game environment.

Patients who are undergoing in-office laryngology procedures (procedures on their vocal cords) will be randomized into a control group augmented reality (AR) group, vibration group, and combined AR and vibration group. The control group will wear a sham augmented reality head set during the procedure. The AR group will have a game played on the head set to distract them during the procedure. The patient will interact with the game use a hand held clicker.

Each participant will answer a survey before and after the procedure assessing their anxiety. Each participant will also wear a one-lead EKG to measure their heart rate through the procedure. The subjective and physiological level will be compared between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing office-based laryngology procedure performed at home institution.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Max pain experienced | measured post-treatment (1 hr).
  Visual analog scale rating of max perceived pain during procedure
Average pain experienced | measured post-treatment (1 hr).
  Visual analog scale rating of average perceived pain during procedure
Pain nervousness experienced | measured post-treatment (1 hr).
  Visual analog scale rating of how nervous about pain patient was during procedure
Time spent thinking about pain | measured post-treatment (1 hr).
  Visual analog scale rating of percent of time spent thinking about pain during procedure
Change in heart rate variability during procedure | calculated post-treatment (1 hr).
  Difference between heart rate variability during procedure compared with pre-procedure
Change in maximum heart rate | calculated post-treatment (1 hr).
  Difference between maximum heart rate during procedure compared with pre-procedure
Change in average heart rate | calculated post-treatment (1 hr).
  Difference between average heart rate during procedure compared with pre-procedure

SECONDARY OUTCOMES:
Change is STAI score | calculated post-procedure (1 hr).
  Measure change in Stait-Trait anxiety inventory State 5 question score pre and post-procedure.
Pain catastrophizing score | calculated pre-procedure (1 hr).
  Pain catastrophizing score
Patient satisfaction | measured post-treatment (1 hr).
  Likert scale rating of satisfaction of treatment group

CONTACTS AND LOCATIONS:
Overall Officials: James J Daniero, MD, Principal Investigator — University of Virginia
Locations (1):
- UVA Fontaine Research Park Building 415, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no intention to share individual participant data with other researchers.

REFERENCES:
- [Background] McCarthy M. US health-care system faces cost and insurance crises. Rising costs, growing numbers of uninsured, and quality gaps trouble world's most expensive health-care system. Lancet. 2003 Aug 2;362(9381):375. doi: 10.1016/s0140-6736(03)14057-3. No abstract available. PMID 12907006
- [Background] Rice T, Rosenau P, Unruh LY, Barnes AJ, Saltman RB, van Ginneken E. United States of America: health system review. Health Syst Transit. 2013;15(3):1-431. PMID 24025796
- [Background] Hoffer EP. The American Health Care System Is Broken. Part 7: How Can We Fix It? Am J Med. 2019 Dec;132(12):1381-1385. doi: 10.1016/j.amjmed.2019.10.003. Epub 2019 Oct 24. PMID 31668898
- [Background] Young S, Shapiro FE, Urman RD. Office-based surgery and patient outcomes. Curr Opin Anaesthesiol. 2018 Dec;31(6):707-712. doi: 10.1097/ACO.0000000000000655. PMID 30148715
- [Background] Saini AT, Citardi MJ, Yao WC, Luong AU. Office-Based Sinus Surgery. Otolaryngol Clin North Am. 2019 Jun;52(3):473-483. doi: 10.1016/j.otc.2019.02.003. Epub 2019 Mar 22. PMID 30905564
- [Background] Shah PD. Patient Safety and Quality for Office-Based Procedures in Otolaryngology. Otolaryngol Clin North Am. 2019 Feb;52(1):89-102. doi: 10.1016/j.otc.2018.08.015. Epub 2018 Sep 22. PMID 30249445
- [Background] Braz J, Solorzano C, Wang X, Basbaum AI. Transmitting pain and itch messages: a contemporary view of the spinal cord circuits that generate gate control. Neuron. 2014 May 7;82(3):522-36. doi: 10.1016/j.neuron.2014.01.018. PMID 24811377
- [Background] Treede RD. Gain control mechanisms in the nociceptive system. Pain. 2016 Jun;157(6):1199-1204. doi: 10.1097/j.pain.0000000000000499. PMID 26817644
- [Background] Zhang Y, Liu S, Zhang YQ, Goulding M, Wang YQ, Ma Q. Timing Mechanisms Underlying Gate Control by Feedforward Inhibition. Neuron. 2018 Sep 5;99(5):941-955.e4. doi: 10.1016/j.neuron.2018.07.026. Epub 2018 Aug 16. PMID 30122375
- [Background] Smith KC, Comite SL, Balasubramanian S, Carver A, Liu JF. Vibration anesthesia: a noninvasive method of reducing discomfort prior to dermatologic procedures. Dermatol Online J. 2004 Oct 15;10(2):1. PMID 15530291
- [Background] Mally P, Czyz CN, Chan NJ, Wulc AE. Vibration anesthesia for the reduction of pain with facial dermal filler injections. Aesthetic Plast Surg. 2014 Apr;38(2):413-8. doi: 10.1007/s00266-013-0264-4. Epub 2014 Jan 24. PMID 24464122
- [Background] Sharma P, Czyz CN, Wulc AE. Investigating the efficacy of vibration anesthesia to reduce pain from cosmetic botulinum toxin injections. Aesthet Surg J. 2011 Nov;31(8):966-71. doi: 10.1177/1090820X11422809. Epub 2011 Oct 14. PMID 22001341
- [Background] Legrain V, Damme SV, Eccleston C, Davis KD, Seminowicz DA, Crombez G. A neurocognitive model of attention to pain: behavioral and neuroimaging evidence. Pain. 2009 Aug;144(3):230-232. doi: 10.1016/j.pain.2009.03.020. Epub 2009 Apr 18. No abstract available. PMID 19376654